CLINICAL TRIAL: NCT06936735
Title: A Phase I Clinical Study Evaluating Safety, Tolerability, Pharmacokinetics and Efficacy of Intravenous HS-20108 in Participants With Advanced Solid Tumors
Brief Title: Phase I Study of HS-20108 in Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20108-101
Record Dates: First submitted 2025-04-14; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor
Keywords: small cell lung cancer; neuroendocrine carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-20108 Ia (Experimental): Phase Ia Dose Escalation
  Interventions: Drug: HS-20108 Monotherapy
- HS-20108 Ib Cohort1 (Experimental): Phase Ib Dose Expansion Cohort 1: Participants with small cell lung cancer will receive varying doses of HS-20108
  Interventions: Drug: HS-20108 Monotherapy
- HS-20108 Ib Cohort2 (Experimental): Phase Ib Dose Expansion Cohort 2: Participants with neuroendocrine carcinoma will receive varying doses of HS-20108
  Interventions: Drug: HS-20108 Monotherapy
- HS-20108 Ib Cohort3 (Experimental): Phase Ib Dose Expansion Cohort 3: Participants with other advanced solid tumors will receive varying doses of HS-20108
  Interventions: Drug: HS-20108 Monotherapy

INTERVENTIONS:
Drug: HS-20108 Monotherapy — Intravenous (IV) Infusion

SUMMARY:
This is a Phase I clinical study of HS-20108. The purpose of this study is to evaluate the safety, tolerability, PK and efficacy of intravenous HS-20108 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase I clinical study to evaluate the safety, tolerability, PK and efficacy of intravenous HS-20108 in patients with advanced solid tumors. The study consists of Phase Ia (dose escalation) and Phase Ib (dose expansion). In Phase Ia, dose escalation will conduct to identify the maximum tolerated dose (MTD) in patients with advanced solid tumors. In Phase Ib, potential indications (such as small cell lung cancer or neuroendocrine carcinoma) will be selected for the early proof-of-concept study of HS-20108 at different doses based on the study data from Phase Ia, the translational medicine research data and R&D progress in the field.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years.
2. Participants with pathologically confirmed advanced solid tumors.
3. At least one measurable lesion in accordance with RECIST 1.1
4. Fresh or archival tumor tissue available for submission.
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0~1.
6. Estimated life expectancy >12 weeks.
7. Reproductive-age women agree to use adequate contraception and cannot breastfeed while participating in this study and for a period of 6 months after the last dose. Likewise, men also consent to use adequate contraceptive method within the same time limit.
8. Females must have evidence of non-childbearing potential.
9. Signed and dated Informed Consent Form.

Exclusion Criteria:

1. Treatment with any of the following:

   Having received cytotoxic chemotherapy agents, investigational drugs, Chinese medicine treatment with anti-tumor indications, or other anti-tumor therapy (including endocrine therapy, molecular targeted therapy, or biotherapy) within 14 days before the first dose of study treatment.

   Having received macromolecular anti-tumor drug therapy (including immunotherapy, such as monoclonal antibody drugs and bispecific antibody drugs) within 28 days before the first dose of study treatment.

   Local radiotherapy for palliation within 2 weeks of the first dose of study drug, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks of the first dose.

   Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) within 4 weeks of the first dose of study drug.
2. Inadequate bone marrow reserve or serious organ dysfunction.
3. Uncontrolled pleural effusion or ascites or pericardial effusion.
4. Known and untreated, or active central nervous system metastases.
5. Active autoimmune diseases or active infectious disease
6. Known to have interstitial pneumonia or immune pneumonia
7. History of severe allergic reaction, serious transfusion reactions or Allergy to any component of HS-20108
8. The subject who is unlikely to comply with study procedures, restrictions, or requirements judged by the investigator.
9. The subject whose safety cannot be ensured or study assessments would be interfered judged by the investigator.
10. Pregnant women, breastfeeding women or woman who has a child-bearing plan during the study.
11. History of neuropathy or mental disorders, including epilepsy and dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2025-04-17 (Estimated); Primary Completion 2027-10-28 (Estimated); Study Completion 2027-11-27 (Estimated)

PRIMARY OUTCOMES:
MTD or MAD of HS-20108 | up to approximately 48 months
  the maximum tolerated dose or maximum appropriate dose

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | up to approximately 48 months
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered an investigational product, which may present with symptoms, signs, disease, or laboratory abnormalities, but do not necessarily have a causality with the investigational product.
Objective response rate (ORR) assessed by investigator | up to approximately 48 months.
  ORR is defined as the percentage of patients with a CR or PR that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.
Disease Control Rate (DCR) | up to approximately 48 months.
  Disease control was deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 5 weeks).
Duration of response (DOR) | up to approximately 48 months.
  Duration of response assessed by RECIST 1.1. Duration of response was defined as the time from when the criteria for CR or PR were first met to the occurrence of an objective disease progression (PD) or death.
Progression-free survival (PFS) | up to approximately 48 months.
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival. Progression-free survival was deﬁned as the time from date of ﬁrst dose until the documentation of objective PD or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.
overall survival (OS) | up to approximately 48 months.
  OS is defined as time from first study treatment to death due to any cause.
Observed maximum plasma concentration (Cmax) of HS-20108 | up to approximately 48 months.
  Cmax of HS-20108
Area Under the Plasma Concentration-Time Curve (AUC) of HS-20108 | up to approximately 48 months.
  AUC of HS-20108

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, BMed, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Jilin Cancer Hospital, Jilin, Jilin, China